CLINICAL TRIAL: NCT04868773
Title: A Phase 1 Study of the Combination of Cabozantinib With Trifluridine/Tipiracil (TAS-102) in Patients With Metastatic Colorectal Adenocarcinoma (mCRC)
Brief Title: Study of Cabozantinib Plus TAS102 in mCRC as Salvage Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Farshid Dayyani, Professor of Clinical Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20216481; UCI 20-134 (Other: CFCCC)
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Metastatic Cancer; CRC
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — cabozantinib; trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: This study is an open-label, single arm clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib in Combination with TAS-102 (trifluridine/tipiracil) (Experimental): Subjects will receive cabozantinib in combination with TAS-102. Patients will receive cabozantinib on Days 1 - 28 and TAS-102 on Days 1-5 and Days 8-12, for a cycle length of 28 days.
  Interventions: Drug: Cabozantinib; Drug: TAS-102

INTERVENTIONS:
Drug: Cabozantinib — Oral cabozantinib
  Other Names: CABOMETYX®; COMETRIQ
Drug: TAS-102 — Oral TAS-102 (trifluridine and tipiracil)
  Other Names: trifluridine and tipiracil

SUMMARY:
This is a phase I clinical trial assessing the safety and recommended phase II dose of cabozantinib in combination with trifluridine/tipiracil (TAS102) in patients with metastatic colorectal carcinoma (mCRC).

DETAILED DESCRIPTION:
Patients with histologically proven colorectal adenocarcinoma not amenable to curative treatment will be eligible to participate for this study. After meeting the eligibility criteria, patients will be given a IP regimen consisting of cabozantinib 20 - 40 mg given orally everyday for 28 days, trifluridine/tipiracil (TAS102) 25 - 35 mg/m2 on Days 1 - 5 and Days 8 - 12 every 28 days, and peg-filgrastim 6 mg subcutaneously on Day 13 every 28 days. Tumor assessments will be completed by CT/MRI every 8 weeks during the first year of treatment and every 3 months after the first year until patient comes off treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed colorectal adenocarcinoma
* Must have locally advanced, recurrent, or metastatic disease not amenable to curative intent surgery or radiation.
* Must have progressed, or not tolerated, a fluoropyrimidine, irinotecan, oxaliplatin, and cetuximab or panitumumab (only for RAS wild-type). Prior exposure to bevacizumab or ramucirumab is allowed. Patients who have exhausted all other standard of care options are also eligible.
* Age ≥ 18 years
* Performance status: ECOG performance status ≤2 (Appendix A).
* Life expectancy of greater than 3 months
* Adequate organ and marrow function as defined below:

  1. leukocytes ≥ 3,000/mcL
  2. absolute neutrophil count ≥ 1,500/mcL
  3. platelets ≥ 100,000/mcl
  4. total bilirubin within normal institutional limits
  5. AST(SGOT)/ALT(SPGT) ≤ 3 X institutional upper limit of normal or ≤ 5 X if liver metastases are present
  6. creatinine <1.5 ULN
  7. hemoglobin ≥ 8 g/dL
  8. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg
  9. (PT)/INR or partial thromboplastin time (PTT) test < 1.3 x ULN
* The effects of cabozantinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  1. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to swallow tablets
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients who have chemotherapy within 2 weeks prior to entering the study
* All toxicities attributed to prior anti-cancer therapy other than alopecia must have resolved to grade 1 or baseline
* Patients may not be receiving any other investigational agents.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102, cabozantinib or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, the following conditions:

  1. ongoing or active infection
  2. Cardiovascular disorders: Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias; uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment; Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose. Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #3.2.8) for at least 1 week before first dose of study treatment.
  3. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
  4. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
  5. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
  6. Lesions invading any major blood vessels. Subjects with lesions invading the intrahepatic vasculature, including portal vein, hepatic vein, and hepatic artery, are eligible.
  7. Other clinically significant disorders that would preclude safe study participation:

  <!-- -->

  1. Active infection requiring systemic treatment (based on investigator assessment). Acute or chronic hepatitis B or C infection, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection.
  2. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
  3. Serious non-healing wound/ulcer/bone fracture
  4. Malabsorption syndrome
  5. Uncompensated/symptomatic hypothyroidism
  6. Moderate to severe hepatic impairment (Child-Pugh B or C)
  7. Requirement for hemodialysis or peritoneal dialysis
  8. History of solid organ or allogenic stem cell transplant
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.5 x the laboratory ULN within 7 days before the first dose of study treatment.
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Prior treatment with cabozantinib
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment. Furthermore, subjects with a history of additional risk factors for torsades de pointes (e.g., long QT syndrome) are also excluded. Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.

Corrected QT (QTc) = QT / ∛RR QT: duration of QT interval RR: duration of RR interval

* History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ.
* Inability to comply with study and follow-up procedures as judged by the Investigator
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Has received a live vaccine within 30 days prior to the first dose of study intervention.
* Has severe hypersensitivity (Grade ≥ 3) to TAS-102 or cabozantinib and/or any of their excipients.
* Has a history or current evidence of any condition (eg, known deficiency of the enzyme dihydropyrimidine dehydrogenase), therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Pregnant or lactating females.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity [DLT] | From the start date of treatment until 4 weeks after the last patient has started treatment, an average of 1 year.
  To determine the Dose Limiting Toxicity (DLT) at Cycle 1 Day 28. A DLT is defined as the occurrence of specific toxicities within the DLT treatment period if judged by the Investigator to be possibly, probably, or definitely related to cabozantinib or TAS-102.
Recommended Phase 2 Dose [RP2D] | From the start date of treatment until 4 weeks after the last patient has started treatment, an average of 1 year.
  To determine the recommended Phase 2 Dose (RP2D) of cabozantinib in combination with TAS-102 in patients with metastatic colorectal carcinoma (mCRC) based on a 3+3 study design.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the start date of treatment until 4 weeks after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  To evaluate the tolerability of administering cabozantinib in combination with TAS-102 in patients with metastatic colorectal cancer from the start of treatment, duration of treatment and up to 4 weeks after completion of study treatment. Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.
Progression-Free Survival of Patients who Received Cabozantinib with TAS-102 | From the start date of treatment until 4 weeks after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall Survival of Patients who Received Cabozantinib with TAS-102 | From date of registration for up to 18 months after last patient is enrolled or until death from any cause, whichever came first
  To evaluate overall survival in patients with metastatic colorectal cancer receiving cabozantinib in combination with TAS-102.
Number of Participants with Objective Response Rate | From the start date of treatment until 4 weeks after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  The ORR is determined by Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) in patients with measurable disease, progression-free, safety regardless of grade and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Dayyani, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

REFERENCES:
- [Derived] Dayyani F, Balangue J, Valerin J, Keating MJ, Zell JA, Taylor TH, Cho MT. A Phase 1 Study of Cabozantinib and Trifluridine/Tipiracil in Metastatic Colorectal Adenocarcinoma. Clin Colorectal Cancer. 2024 Mar;23(1):67-72. doi: 10.1016/j.clcc.2023.11.001. Epub 2023 Nov 27. PMID 38103947